CLINICAL TRIAL: NCT01245868
Title: Spinal Anaesthesia for Knee Arthroscopy: Does Lignocaine Shorten the Effect of Bupivacaine?
Brief Title: Spinal Anaesthesia for Knee Arthroscopy: Does Lignocaine Shorten the Effect of Bupivacaine
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Frederikssunds Hospital, Denmark (Other)
Responsible Party: Principal Investigator, Jon Jacobsen, Chief consultant, Frederikssunds Hospital, Denmark
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: FRS-AN2009-03-09
Record Dates: First submitted 2010-06-14; First posted 2010-11-23 (Estimated); Last update posted 2015-05-08 (Estimated); Status verified 2015-05

CONDITIONS: Spinal Anesthesia
Keywords: Spinal anaesthesia; Bupivacaine; Lidocaine; Duration of blockade
MeSH Terms: interventions — Lidocaine; Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Bupivacaine (Experimental): Bupivacaine as used routinely
  Interventions: Drug: bupivacaine
- Lidocaine added to bupivacaine (Placebo Comparator): lidocaine is added to bupivacaine
  Interventions: Drug: Lidocaine; Drug: bupivacaine

INTERVENTIONS:
Drug: Lidocaine
  Arms: Lidocaine added to bupivacaine
Drug: bupivacaine

SUMMARY:
The purpose of the study is to investigate if a small amount of lignocaine added to bupivacaine for spinal anesthesia to patients planned for arthroscopic knee surgery, can shorten the duration of the sensoric and the motoric blockade.

ELIGIBILITY:
Inclusion Criteria:

* The patient want spinal anaesthesia
* No contradictions against spinal anaesthesia
* Healthy people (ASA-score 1 or 2)
* Body mass index < 35 and between 155 and 190 cm

Exclusion Criteria:

* Known allergic reactions to planned drugs
* Neurologic disturbances
* Diabetes

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2009-11; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Duration of spinal blockade | Repeating monitoring every 15 minutes after applying the blockade, up to 360 minutes.

SECONDARY OUTCOMES:
Time to fulfillment of discharge criteria from the hospital. | Evaluated every 15 minutes after the operation up to 360 minutes. On average 200 to 300 minutes.

CONTACTS AND LOCATIONS:
Overall Officials: Jon Jacobsen, M.D., Principal Investigator — Frederikssunds Hospital, Denmark
Locations (2):
- Denmark (2):
  - Dep. of anesthesiology, Hospital of Frederikssund, Frederikssund
  - Jon Jacobsen, Frederikssund